CLINICAL TRIAL: NCT06273332
Title: Assessment of the AI-assisted Registration Versus Conventional Point-based Registration on CBCTs With Heavy Metal Artifacts
Brief Title: Assessment of the Artifical Intelligence Assisted Registration Versus Conventional Point Based Registration on Cone Beam-computed Tomography (CBCT) With Heavy Metal Artifacts
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nehal Ibrahim Ahmed Shobair, principal investigator, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AI surgery protocol
Record Dates: First submitted 2024-02-05; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Registration Accuracy
Keywords: Point-based registration; AI registration; Accuracy; Digital implant planning

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-assisted registration (Experimental): 3D model registration will be carried out using artificial intelligence
  Interventions: Other: AI-assisted registration
- Point-based registration (Active Comparator): 3D model registration will be carried out using point-based approach
  Interventions: Other: Point-based registration

INTERVENTIONS:
Other: AI-assisted registration — We will use artificial intelligence to register 3d model on intra-oral scan
  Arms: AI-assisted registration
Other: Point-based registration — We will use five references points or more to perform model registration
  Arms: Point-based registration

SUMMARY:
Our study investigates the accuracy and duration needed for 3D model registration using artifical intelligence (AI) assistance compared to conventional point-based registration. Manual segmentation of all cone beam computed tomography (CBCT) scans will be performed before the registration procedure.

DETAILED DESCRIPTION:
CBCT images and intraoral scans will be screened following specific eligibility criteria. 16 CBCT images and intraoral scans that will meet the inclusion criteria will undergo manual segmentation via 3D medical image processing software. Afterward, point-based registration and AI-assisted registration will be performed by a single operator using specialized implant planning software. Then, the registration accuracy will be examined by measuring the distances between the three-dimensional models of CBCT data and intraoral scans. Also, the duration required for registration will be calibrated and recorded by a stopwatch.

ELIGIBILITY:
Inclusion Criteria:

CBCT scans for either the maxilla or mandible or both and intraoral scans or manual impressions with metal restorations.

Exclusion Criteria:

Scans without metal restorations.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-02-25 (Estimated)

PRIMARY OUTCOMES:
Registration accuracy | immediately after the procedure
  Distance between registered 3d model and CBCT in millimeters

SECONDARY OUTCOMES:
Duration for registration | During the procedure
  time taken for registration procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Private maxillofacial digital lab, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
no data will be shared